CLINICAL TRIAL: NCT06404866
Title: Satisfaction With eMotion in a Diverse Group of Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kelly L. Wierenga, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19153
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Events; Emotions
Keywords: Emotion Regulation
MeSH Terms: conditions — Cardiovascular Diseases; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- eMotion Intervention (Experimental): This is a single-group study assessing participation satisfaction with the 10-week eMotion intervention. The eMotion intervention is based on feasibility testing of the successful in-person program with critical refinement to improve accessibility. eMotion has undergone subsequent content validity testing with intervention development, self-management, cardiovascular health, and health information technology delivery experts. eMotion teaches a carefully selected repertoire of emotion regulation strategies well suited for adults following a first cardiac event.
  Interventions: Behavioral: eMotion

INTERVENTIONS:
Behavioral: eMotion — Participants will complete one lesson per week. The weekly education is targeted to women and contains personalized content via a variety of diverse lesson narratives. Each week participants listen to scripted sessions they can complete on their own time regarding each of the weekly topics (lasting about 30 minutes). At the end of the week, they then meet individually with a study team member virtually to discuss the same subject.

SUMMARY:
The eMotion intervention, developed by the PI, provides training on multiple emotion regulation skills based on leading theories and evidence-based emotion regulation interventions. After initial pilot testing of eMotion, the investigators revised the intervention to make it more relevant to women from diverse backgrounds, as these women are disproportionately impacted by social determinants of health that complicate their recovery. It is important to revise the intervention to be acceptable to women from diverse backgrounds and to address their unique needs. The investigators want to explore if women from diverse backgrounds find the revised intervention relevant, meaningful, and easy to understand and apply to their lives. Their feedback will help investigators further revise the intervention to make it acceptable for this population.

DETAILED DESCRIPTION:
This is a single-group study assessing participation satisfaction with the 10-week eMotion intervention. The eMotion intervention is based on feasibility testing of the successful in-person program with critical refinement to improve accessibility. eMotion has undergone subsequent content validity testing with intervention development, self-management, cardiovascular health, and health information technology delivery experts. eMotion teaches a carefully selected repertoire of emotion regulation strategies well suited for adults following a first cardiac event.

Participants will complete one lesson per week. The weekly education targets women and contains personalized content via diverse lesson narratives. Each week, participants listen to scripted sessions they can complete on their own time regarding each weekly topic (lasting about 30 minutes). At the end of the week, participants meet individually with a study team member virtually to discuss the same subject. The lessons will be comprised of rich emotion regulation strategies selected based on the efficacy and preferences of middle-aged and older adults. The 10 lessons covered are, 1) safe exercise guidelines and strategies, 2) why emotions matter and identifying emotions, 3) becoming an emotion detective, 4) mindful walking, 5) selecting and changing situations, 6) evaluating a challenge and responding, 7) choosing what to pay attention to, 8) thinking positively, 9) emotional responses for change, and 10) changing strategies and recognizing strengths.

Baseline and concluding surveys will be completed by participants that will take approximately 20 minutes. The baseline and concluding measures will help investigators characterize our sample and further understand risk factors that may contribute to dissatisfaction or confusion. After each week's lessons, each participant will be sent an individualized survey link to complete an IU RedCap survey with questions covering participant satisfaction with the eMotion intervention. The intervening surveys (weeks 2-9) should take approximately 10 minutes to complete each week.

Each week's content, including lessons, and surveys will last approximately 45-60 minutes, or 10 hours across the entire intervention period.

ELIGIBILITY:
Inclusion Criteria:

* First-time major cardiac event as documented in the medical record
* Lives independently
* Has at least mild symptoms of depression (determined by Patient Health Questionnaire-8 [PHQ-8] scores of 5 or greater) and/or at least mild symptoms of anxiety (determined by the General Anxiety Disorder [GAD-7] scores of 5 or greater).

Exclusion Criteria:

* Does not understand both spoken and written English
* In palliative care or hospice
* Legally blind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible if self-identifies as a woman
Enrollment: 5 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Distress-Depression and Anxiety Stress Scale | three months
  Changes in the level of distress over time. The minimum value (Normal):0 The maximum value (extremely severe): 42 Higher scores equate to worse outcome.

SECONDARY OUTCOMES:
Physical Activity | three months
  Change in amount of time exercising at moderate or greater intensity

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Wierenga, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No